CLINICAL TRIAL: NCT04753073
Title: Treatment of Cervical Intraepithelial Neoplasia (CIN) Grade III With Non-invasive Physical Plasma
Acronym: ZGynO_CINIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZGynO_CIN_III
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Cervical Intraepithelial Neoplasia III
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIPP (Experimental): Treatment of the NIPP group with physical low-temperature plasma, subsequently within 8 weeks LEEP-Exzision
  Interventions: Procedure: Non-invasive physical plasma
- Controll (No Intervention): LEEP-Exzision

INTERVENTIONS:
Procedure: Non-invasive physical plasma — Treatment with non invasive physical low-temperature plasma
  Arms: NIPP

SUMMARY:
The aim of the prospective, unicenter proof-of-principle study is to investigate the anti-neoplastic effectiveness of NIPP against CIN III lesions.

* The aim of this project is to evaluate the potential of a previous NIPP treatment to significantly reduce the invasiveness of the LEEP excision.
* Another aim of this study is to investigate cellular / molecular effects of NIPP following the in-vivo treatment of the cervix using molecular biological methods. For this purpose, tissue treated with plasma is taken after defined periods of time by mini biopsy and examined using molecular biological, histological and microscopic methods.

DETAILED DESCRIPTION:
Cervical intraepithelial neoplasms (CIN), classified into severity levels CIN I to III, can be precursors to cervical cancer (CC), the world's third most common cancer in women (270,000 deaths / year), which radical therapies are often associated with lifelong severe physical and emotional stress. Cross-sectional studies found a prevalence for CIN of 62 per 1,000 women and incidences of 1.2 (CIN I), 0.8 (CIN II) and 0.7 (CIN III) per 1,000 women per year (highest incidence of CIN between 20 and 24 years) age). The standard therapy for the treatment of CIN III by LEEP excision is associated with an increase in mortality of 17%. CIN III, in particular, is associated with a significant decline in quality of life, psychological well-being and sexual health, although on average only about 12% of CIN III lesions progress to invasive CC. The resulting over-treatment (in around 8-9 out of 10 patients) with invasive procedures is a serious problem for affected women, health care providers and the health economy.

The NIPP treatment is a tissue-sparing, pain-free, easy to carry out and outpatient treatment method without anesthesia and hospitalization. A non-randomized, one-arm feasibility study at the Department of Women's Health (649 / 2017BO1) already showed the effectiveness of a NIPP treatment.

Clinical implications for CIN III:

* A previous NIPP treatment should significantly reduce the invasiveness of the LEEP excision.
* If the oncological safety of NIPP treatment is comparable (histological complete remission of CIN III), NIPP is to be established as a safe alternative to LEEP excision in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

  * Histologically confirmed CIN III
  * Clearly visible transformation zone of the portio and margins of the lesions according to T1 / T2
  * signed written consent

Exclusion Criteria:

* Not fully visible transformation zone

  * Indication of an invasive disease
  * Serious cardiovascular diseases
  * Patients who only want to undergo a LEEP excision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of histological complete remission | 8 Weeks
  Rate of histological complete remission of the CIN III at the time of the LEEP excision

SECONDARY OUTCOMES:
Rate of partial histological remission | 8 Weeks
  Rate of partial histological remission of the CIN I / II
Rate of decreased HPV viral load | 8 Weeks
  Rate of decreased HPV viral load in tissues
Pain and quality of life | 8 Weeks
  Pain and quality of life (Freiburg index for patient satisfaction)
  1. Pain assessment i) previous to, ii) during, iii) 4 h after, iv) 2 days after, v) 1 week after NIPP treatment, min/max values: 0 - 10, higher scores mean worse outcome
  2. Satisfaction assessment, min/max values: 1-6, higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weiss, Dr. med.q, Principal Investigator — Department of Women's Health, University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Department of Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henes M, Matovina S, Rottscholl R, Feng YS, Fleischhacker A, Wang G, Enderle M, Awakowicz P, Brucker SY, Weiss M. Tissue preserving non-invasive physical plasma treatment for cervical squamous intraepithelial neoplasia grade 3-a prospective randomized, controlled clinical trial. Front Med (Lausanne). 2025 Nov 7;12:1669933. doi: 10.3389/fmed.2025.1669933. eCollection 2025. PMID 41282018